CLINICAL TRIAL: NCT06538389
Title: High Cannabidiol (CBD) Standardized Extract for Aromatase Inhibitor-Induced Arthralgia - A Randomized Controlled Double Blind Clinical Trial
Brief Title: High Cannabidiol Plant Extract (BRC-001) to Improve Aromatase Inhibitor-Induced Arthralgia in Women With Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Biopharmaceutical Research Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23710; NCI-2024-05417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23710 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-07-16; First posted 2024-08-05 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Breast Adenocarcinoma; Breast Ductal Carcinoma In Situ; Estrogen Receptor-Positive Breast Carcinoma; Progesterone Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Specimen Handling; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (BRC-001) (Experimental): Participants will be started on a flexible dosing regimen of BC-001, initiating therapy at 200 mg daily and up-titrated based on tolerability over 2 weeks to a maximum of 800 mg daily. Dose increases are recommended to take place in the evening, beginning the evening dose of Day 2. During the Titration Period, study participants may increase the study agent dose every 2 days by 1 mL total (.5 mL per dose) as tolerated. The increment of increase for BRC-001 is 100 mg per 1.0 mL. Patients receive BRC-001 PO BID for up to 3 months. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: BRC-001; Other: Questionnaire Administration
- Arm II (Placebo) (Placebo Comparator): Placebo will be self-administered with twice daily doses according to the Titration Period schedule for the first two weeks to the highest tolerable dose up to 4 mL twice daily. Patients receive placebo PO BID for up to 3 months. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: BRC-001 — Given PO
  Other Names: Cannabidiol; CBD; CBD Oil
  Arms: Arm I (BRC-001)
Drug: Placebo Administration — Given PO
  Arms: Arm II (Placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests the effectiveness of cannabidiol (CBD) plant extract (BRC-001) in improving joint stiffness and pain (arthralgia) in women with breast cancer taking aromatase inhibitors (AIs). AIs lower blood levels of estrogen in postmenopausal women to reduce breast cancer recurrence. Women on AI therapy may experience joint stiffness, pain and arthritis symptoms as a side effect of the medication. Some women stop AI therapy due to these side effects and do not receive the maximum benefit from the medication. CBD is derived from the same plant family as marijuana but is not associated with a "high" or mind-altering effect and is not habit-forming. Research in animals and humans indicates that CBD might decrease inflammation in joint tissues and may help reduce chronic pain in ailments such as arthritis. BRC-001 may reduce joint pain in women with breast cancer taking AIs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the preliminary efficacy of BRC-001 versus placebo by change in Brief Pain Inventory-Short Form (BPI-SF) worst pain severity scores from 0 to 3 months.

SECONDARY OBJECTIVES:

I. To evaluate indicators of preliminary efficacy of BRC-001 on joint symptoms of pain and stiffness assessed by BPI-SF total pain severity and total pain interference scores and Visual Analog Scale-Pain.

II. To evaluate tolerability by adverse events, anxiety by Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short Form (SF) 6a, sleep by PROMIS Sleep Disturbance SF 4a, quality of life by Functional Assessment of Cancer Therapy-Endocrine System (FACT-ES).

III. To evaluate safety by clinical laboratory tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin).

IV. To evaluate changes in physical function by dynamometer measurements of grip strength.

EXPLORATORY OBJECTIVES:

I. To evaluate blood-based biomarkers related to aromatase inhibitor-induced arthralgia (AIIA) and BRC-001 versus (vs) placebo.

II. Pharmacokinetics of BRC-001.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive BRC-001 orally (PO) twice daily (BID) for up to 3 months. Patients also undergo blood sample collection on study.

ARM II: Patients receive placebo PO BID for up to 3 months. Patients also undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Postmenopausal by last menses > 12 months or medically induced menopause in premenopausal women for AI therapy use
* At least 5 years since other malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or adequately treated stage I or II cancer from which the patient is currently in complete remission
* Ability to read and understand English, Spanish, or translations by interpreters for questionnaires
* Histologically confirmed primary invasive adenocarcinoma of the breast or ductal carcinoma in situ of the breast

  * Stage 0, I, II, or IIIA disease
  * No metastatic disease
* Must have undergone definitive breast cancer surgery and recovered
* Must have completed adjuvant chemotherapy as applicable, including systemic chemotherapy, anti-HER2 therapy, and/or radiation therapy
* Estrogen-receptor positive (ER+) and/or progesterone-receptor positive (PR+)
* Currently taking a third-generation aromatase inhibitor (AI) (e.g., anastrozole [Arimidex (registered trademark)], letrozole [Femara (registered trademark)], or exemestane [Aromasin (registered trademark)]) for ≥ 90 days prior to registration with plans to continue for ≥ 180 days after registration
* Must have a worst pain/stiffness of ≥ 4 on the Brief Pain Inventory (BPI) (item #2) that has started or increased with AI therapy

Exclusion Criteria:

* < 3 months since prior cannabinoid containing cannabis or hemp products including CBD, tetrahydrocannabinol (THC), Marinol, and Epidiolex and must agree to refrain from use from sources outside of this study
* < 28 days since prior investigational agents
* Medical therapy, alternative therapy, or physical therapy for joint pain/stiffness within the past 30 days
* Narcotic use within 14 days of registration
* Patients may have received corticosteroid treatment; however, the following criteria apply:

  * Patients must not have received oral or intramuscular corticosteroids within 28 days prior to registration
  * Patients must not have received intra-articular steroids to the study, or any other, joint within 28 days prior to registration
* Patients must not have received topical analgesics (e.g., capsaicin preparations) to the study joint or any other analgesics (e.g., opiates, tramadol; with exception of nonsteroidal anti-inflammatory drugs [NSAIDs] and acetaminophen) within 14 days prior to registration
* History of bone fracture or surgery of the afflicted hands, knees, and/or other joints within 6 months prior to registration
* Any uncontrolled illness including ongoing or active infection
* Known allergies or contraindications to cannabis
* Significantly impaired hepatic function (alanine aminotransferase [ALT] > 5 x upper limit of normal [ULN] or total bilirubin [TBL] > 2 x ULN) OR the ALT or aspartate aminotransferase (AST) > 3 x ULN and TBL > 2 x ULN (or international normalized ratio [INR] > 1.5
* Grade 3+ renal impairment
* Clinically significant lab abnormalities in ALT, AST, total bilirubin, hemoglobin, hematocrit, or creatinine or any other laboratory tests that in the opinion of the investigator would prevent the patient from safely participating in the study
* Having current thoughts of suicide or self-harm or history of suicidal ideation or attempted suicide
* Meeting Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria for current major psychiatric illness, such as bipolar disorder, major depression, or psychosis (including schizophrenia and affective psychosis)
* History of seizure disorder
* Concomitant administration with drugs that may interact adversely with CBD including warfarin, theophylline, amiodarone, anti-epileptic (e.g., clobazam, stiripentol, valproate, topiramate), anticonvulsant (e.g., diazepam, lamotrigine, phenytoin, ethosuximide, oxcarbazepine, pregabalin, tigabine, gabapentin); 3) barbiturate (e.g., phenobarbital, hexobarbital), benzodiazepine (e.g, chlordiazepoxide, clonazepam), opioid/narcotic (e.g, codeine, morphine)
* Concomitant administration of cyclin-dependent kinase 4/6 inhibitors, such as abemaciclib, with AI therapy
* Following a physical examination, the patient has any abnormalities that, in the opinion of the investigator would prevent the patient from safely participating in the study
* Other active malignancy
* Any other condition or medication use that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Participants unwilling to abstain from donation of blood during the study
* Participants who plan to travel outside of the United States during the study period
* Women with childbearing potential are not eligible to participate. The study is for postmenopausal women taking aromatase inhibitors for adjuvant endocrine therapy
* Participants with cognitive impairment are excluded due to dose titration instructions and completion of questionnaires
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Brief Pain Inventory-Short Form (BPI-SF) score | From 0 to 3 months
  The Brief Pain Inventory (BPI) can assess the severity of chronic and acute pain for both behavioral and pharmacological pain interventions. Higher scores from 0 (no pain) to 10 (pain as bad as you can imagine) indicate increased levels of pain. Changes will be summarized by treatment arm. Data will be represented using means/medians.

SECONDARY OUTCOMES:
Changes in Visual Analog Scale (VAS) for Pain | From 0 to 3 months
  The Visual Analogue Scale (VAS) measures pain intensity with two end points (0=no pain and 10=worst pain). Changes will be summarized by treatment arm. Data will be represented using means/medians.
Changes in Functional Assessment of Cancer Therapy-Endocrine System (FACT-ES) scores | From 0 to 3 months
  FACT-ES Score measures physical, social and family, emotional, and functional well-being and endocrine symptoms. Higher scores reflect better well-being and fewer symptoms. Score range is 0 to 220. Changes will be summarized by treatment arm. Data will be represented using means/medians.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be characterized using the descriptions and grading scales of the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Higher grades indicate greater severity.
Changes in PROMIS Emotional Distress-Anxiety Short Form (SF) 6a Score | From 0 to 3 months
  The Emotional Distress-Anxiety SF consists of 7 questions regarding feelings of distress/anxiety in the past 7 days. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety. Changes will be summarized by treatment arm. Data will be represented using means/medians.
Changes in PROMIS Sleep Disturbance Short Form (SF) 4a Score | From 0 to 3 months
  The Sleep Disturbance SF 4a is an 8-item tool with questions regarding sleep disturbance. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance. Changes will be summarized by treatment arm. Data will be represented using means/medians.
Changes in Physical Function by Grip Strength | At 0 and up to 3 months
  Grip strength will be quantitated by hand dynamometer (Jarman) at 0 and 3 months. The dominant hand will be recorded for each participant at baseline. This test involves squeezing a dynamometer for 2 to 3 seconds and then releasing. Changes will be summarized by treatment arm. Data will be represented using means/medians.
Changes in Alanine Aminotransferase (ALT) | At 0, 1, and 3 months
  Blood samples will be obtained for testing of alanine transaminase (ALT). An increased ALT indicates a sign of liver dysfunction. Changes will be summarized by treatment arm. Data will be represented using means/medians.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Yee, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States